CLINICAL TRIAL: NCT02653300
Title: An Open-Label Pilot Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Potential of Oral Insulin to Reduce Liver Fat Content and Fibrosis in Patients With Nonalcolholic Steatohepatitis (NASH)
Brief Title: A Pilot Study to Assess the Safety of Oral Insulin in Patients With Nonalcolholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORA-D-N01
Record Dates: First submitted 2015-12-24; First posted 2016-01-12 (Estimated); Results first posted 2021-09-23 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH); Type2 Diabetes Mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Insulin (Experimental): treatment
  Interventions: Biological: Oral Insulin

INTERVENTIONS:
Biological: Oral Insulin — all patients will receive treatment regimen of a soft gel capsule of ORMD-0801.

SUMMARY:
This is an open, pilot study using the oral ORMD-0801 insulin formulation in patients with NASH and confirmed type 2 DM or pre-diabetes. The study will consist of a Screening, placebo run-in, treatment phase and end-of-study phase.

DETAILED DESCRIPTION:
This exploratory study will first enroll 10 patients with NASH and type 2 DM, to evaluate the safety of oral insulin and to measure the change in liver fat content.

At the completion of their 4-week follow-up period, results will be presented to the Helsinki Committee. Following approval, an additional 20 patients will be enrolled. The size of the study population was determined by the investigator (with literature review) to be sufficient to show trends of reducing liver fat content by analysis of MRI PDFF (MRI-Proton Density Fat Fraction) images, the FibroMax™ Test and Fibroscan® including Controlled Attenuation Parameter (CAP™). CAP™ is a measure of the ultrasound attenuation to quantify steatosis in the liver.

ELIGIBILITY:
Inclusion Criteria:

* Known type 2 DM according to American Diabetic Association (one of the three needed): Fasting Plasma Glucose ≥126 mg/dl or 2h postprandial (PG) following 75g OGTT ≥ 200 mg/dl or HbA1C > 5.7% or on treatment with metformin
* Abdominal ultrasound (US) proven fatty liver performed within 6 months before randomization, confirmed by central US.
* Fat concentration in the liver of S2 (moderate steatosis, 6-32% hepatocytes with steatosis) or more as measured by Fibromax.
* Signature of the written informed consent.
* Negative pregnancy test at study entry for females of child bearing potential.
* Females must have a negative urine pregnancy test result at screening, prior to the start of the run-in period, and at initiation of active dosing. A negative urine and serum pregnancy test must be obtained prior to active dosing. Males and females of childbearing potential must use two methods of contraception.
* Females of non-childbearing potential are defined as postmenopausal who a) had more than 24 months since last menstrual cycle with menopausal levels of FSH, b) who are surgically menopausal.
* For hypertensive patients, hypertension must be controlled by stable dose of anti-hypertensive medication for at least 2 months prior to screening with BP < 150/<95 mmHg
* Patients previously treated with vitamin E (>400IU/day).
* Glycaemia must be controlled (Glycosylated Hemoglobin A1C ≤9%) while any HbA1C increment should not exceed 1% during 6 months prior to enrolment).

Exclusion Criteria:

* Patients with active (acute or chronic) liver disease other than NASH (e.g. viral hepatitis, genetic hemochromatosis, Wilson disease, alpha 1antitripsin deficiency, alcohol liver disease, drug induced liver disease) at the time of randomization.
* ALT or AST ≥ 2 times ULN
* Abnormal synthetic liver function (serum albumin ≤3.5gm%, INR >1.3).
* Known alcohol and/or any other drug abuse or dependence in the last five years.
* Weight >120 Kg
* Known history or presence of clinically significant cardiovascular, gastrointestinal, metabolic (other than diabetes mellitus), neurologic, pulmonary, endocrine, psychiatric, neoplastic disorder or nephrotic syndrome.
* History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs including bile salt metabolites (e.g. inflammatory bowel disease (IBD), previous intestinal (ileal or colonic) operation, chronic pancreatitis, celiac disease or previous vagotomy.
* Weight loss of more than 5% within 6 months prior to randomization.
* History of bariatric surgery.
* Uncontrolled blood pressure BP ≥150/95.
* Non type 2 DM (type I, endocrinopathy, genetic syndromes etc).
* Patients with HIV.
* Daily alcohol intake >20 g/day for women and >30 g/day for men.
* Treatment anti-diabetic medications other than metformin, such as DPP-4 inhibitors, GLP-1 receptor agonists, TZDs, etc.
* Metformin, Fibrates, Statins, not provided on a stable dose in the last 6 months.
* Patients who are treated with Valproic acid, Tamoxifen, Methotrexate, Amiodaron.
* Chronic treatment with antibiotics (e.g. Rifaximin).
* Homeopathic and/or Alternative treatments.
* Uncontrolled hypothyroidism defined as Thyroid Stimulating Hormone >2X the upper limit of normal (UNLN).
* Patients with renal dysfunction: eGFR< 40 ml/min.
* Unexplained serum creatinine phosphokinase

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rifaat Safadi, M.D., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Ratziu V, Bellentani S, Cortez-Pinto H, Day C, Marchesini G. A position statement on NAFLD/NASH based on the EASL 2009 special conference. J Hepatol. 2010 Aug;53(2):372-84. doi: 10.1016/j.jhep.2010.04.008. Epub 2010 May 7. No abstract available. PMID 20494470
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Lin SC, Heba E, Bettencourt R, Lin GY, Valasek MA, Lunde O, Hamilton G, Sirlin CB, Loomba R. Assessment of treatment response in non-alcoholic steatohepatitis using advanced magnetic resonance imaging. Aliment Pharmacol Ther. 2017 Mar;45(6):844-854. doi: 10.1111/apt.13951. Epub 2017 Jan 24. PMID 28116801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Insulin
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Oral Insulin
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Israel | 10
BMI [Mean (Standard Deviation); unit: Kg/M^2] — Body Mass Index
  Kg/M^2 | 32.08 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in MRI-Proton Density Fat Fraction (MRI-PDFF)
Description: Absolute Change in MRI-Proton Density Fat Fraction (expressed as percent fat in the liver) from baseline to week 12
Time Frame: Two timepoints: Baseline (week 0) and Week 12
Measure: Mean (Standard Deviation); unit: percentage fat in the liver
Arm/Group | Oral Insulin
Number analyzed (Participants) | 8
percentage fat in the liver
  MRPDFF (%) at baseline | 21.3 (7.2)
  MR PDFF (%) at Week 12 | 14.4 (6.3)
  Absolute Mean Change in MR PDFF (%) from Baseline | -6.9 (6.8)
Statistical Analysis 1: Comparison: Oral Insulin; Test type: Other; p = 0.03125, Sign test

2. Secondary Outcome: Mean Transient Elastography Measurement (Fibroscan)
Description: Mean Transient elasticity, measured in kPA (kilo Pascal),
Time Frame: Two timepoints: Baseline (week 0) and Week 12
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Oral Insulin
Number analyzed (Participants) | 8
kPa
  Baseline | 8.6 (1.5)
  Week 12 | 7.4 (2.5)

3. Secondary Outcome: Mean Fibrosis Score CAP™ (FibroMax)
Description: Mean fibrosis score (severity scale of liver fibrosis) measured at baseline and week 12. Fibrosis Score CAP measures the amount of steatosis (fatty change) in the liver. The CAP score is measured in decibels per meter (dB/m). It ranges from 100 to 400 dB/m with higher values indicating more fatty change
Time Frame: Two timepoints: Baseline (week 0) and Week 12
Measure: Mean (Standard Deviation); unit: dB/M
Arm/Group | Oral Insulin
Number analyzed (Participants) | 8
dB/M
  Mean Fibrosis Score at Baseline | 338.5 (15.6)
  Mean Fibrosis Score at week 12 | 315.5 (39.6)

ADVERSE EVENTS:
Time Frame: twelve weeks (Baseline to 12 weeks)
Arm/Group | Oral Insulin
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
This is a pilot study with ten subjects enrolled, and eight subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol: Clinical Protocol ORA-D N01 (2018-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT02653300/Prot_000.pdf